CLINICAL TRIAL: NCT02747745
Title: Theoretical Based Case Management Intervention for Dementia Family Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chien, Chiu, Associate Professor, Chang Gung University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMRPD1F0051; CMRPD1F0051 (Other Grant/Funding Number: Chang Gung Memorial Hospital)
Record Dates: First submitted 2016-04-10; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Dementia
Keywords: Caregivers; Case Management; Community Dwelling
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Group receive no intervention
- Interventional Group (Experimental): Four risk areas reflecting the great needs of FCGs of PWDs: depressive symptoms, burden, distress to problematic behaviors of PWDs and healthy behaviors.
  Interventions: Behavioral: Four risk areas reflecting the great needs of FCGs of PWDs

INTERVENTIONS:
Behavioral: Four risk areas reflecting the great needs of FCGs of PWDs — The intervention involves home visits & phone calls from the case manager to the dyads, and receiving telephone calls from FCGs. The case manager will target the prioritized risk from the 4 risk areas of FCG problems and healthy behaviors. The intervention mainly consists of needs assessment and nursing education on home environment modification and safety, behavioral management and communication skills; home-based cognitive stimulation on PWD with simple mathematical practice, patient preferred leisure activities and reminiscence by old time photos, stories and toys; brief consultation on 4 risk areas related to FCG stress; and case management to refer the dyads to the hospital-based dementia centers and community resources.
  Arms: Interventional Group

SUMMARY:
The growing number of persons with dementia (PWDs) calls for policy changes and service innovation. Recent case management (CM) research is recognized by its positive impacts on family caregivers (FCGs) of PWDs. However, research gaps are identified, including the paucity of theoretical based CM practice and a lack of mediator effects. Therefore, the original purpose of this five-year project was to implement a theoretical-based randomized controlled CM intervention for FCGs of early to moderate PWDs at home based on a stress model and tailor to needs prioritized by FCGs. This project was funded by the Minister of Scientific and Technology for the first two years and accomplished the first two aims: 1. First year: to develop and test the psychometric properties of related instruments and protocol (cross-sectional study); 2. Second year: to conduct a feasibility test for the CM intervention (a pilot RCT). The purpose of the current project is to achieve aim 3 (three years): to implement a 4-month CM intervention (the main RCT). In total, there will be 2 home visits, 2 phone calls to the dyads, and receiving telephone calls from the FCGs during the working hours. Investigator will collect 4-time point data at T0 for base line data, T1 (after the recruitment, 4 th month, the first follow up), T2 (after the recruitment, 6th month, the second follow up) and T3 (after the recruitment,12 th month). Investigator will recruit 76 dyads in three years (38 dyads for each group)(n = 152 in total). The primary outcomes are FCG QoL and PWD behavioral problems, while the secondary outcome is the percentages of PWD status (i.g. nursing home admission) and the frequency of PWD acute hospitalization. Investigator will also test of mediator effect of FCG self efficacy using statistical analysis method such as Hierarchical Linear Modeling (HLM).

DETAILED DESCRIPTION:
The primary care physicians in the memory disorder clinics at the participating hospitals (Chang-Gung Memorial Hospital at Lin-Kuo, Chang-Gung Memorial Hospital-Taoyuan branch, Catholic Mercy Hospital at Hukou, Hsinchu county) will receive a written letter to explain the purpose of this project and the eligible criteria of PWDs and their FCGs. Debriefing can be provided upon request. Then the participating physicians will help to identify eligible dyads; while one trained research assistant (RA) is responsible for CM implementation (RA I), and the second RA (graduate students, RA II) will be responsible for data collection in each time point.

To increase the feasibility of this project, the inclusion criteria of PWDs are made to reflect the recruiting site reality, including: (1) age being older than 60 years old; (2) having a primary FCG or a secondary FCG who can provides sufficient information and assistant for the PWD; co-residence is not required; (3) PWDs are those with cognitive impairment confirmed by the primary or secondary FCG or participating neurologists. The exclusion criteria of PWDs include: (1) acute illnesses, impaired sensory symptoms (hearing loss and severe visual problems); (2) acute agitation which requires emergency treatment; (3) chronic alcohol abuse or use of drugs which possibly affect central nervous system functions; (4) presence of major psychiatric disorders within the last 2 years; (5) neurological or systemic illness (e.g. delirium, hypoxia, or unstable thyroid dysfunction); (6) no primary FCG or secondary FCG.

Investigator will screen for FCGs who report and meet the criteria of moderate levels of severity in the following risk areas (Table 1): depressive symptoms, burden, distress to problematic behaviors of PWDs and healthy behaviors. The definition of primary FCG include: (1) age 18 years old or greater; (2) at least providing the most assistance (4 hours a day) to their relatives with dementia for the past three months or those who conduct secondary care to their relatives, meaning that these FCGs supervise the hired care assistants or foreign helpers who actually take care of the patients; co-residency is not required for family caregivers. Exclusion criteria of family caregivers include: (1) documented cognitive or mental disorder, such as severe memory problems or major affective disorders; (2) hearing or visual impairments which are not properly corrected; (3) prescribed drugs known to impair or enhance attention, e.g., antidepressants, barbiturates, or other depressants, amphetamines; (4) insufficient command of Mandarin, Taiwanese; (5) participation in other interventions which may contaminate the results of this study.

In previous project, the satisfactory level of our case management training course was high. All the trainees had the highest regard toward the professional quality of the content and the instructors (Chiu et al, 2013). One of the case managers served as research assistant in the previous project and will continue to work with us as interventionist upon funded. Investigator will conduct a three-year RCT involving repeated measures at four time points: baseline screening (T0), 4th month (the end of the intervention, T1), 6th month (post-treatment follow up, T2), 12th month (T3).

Randomization Randomization takes place after baseline assessment. An external independent person establishes the random order using random number tables.

CM Intervention Protocol The 4-month CM intervention on FCGs of PWDs involves 2 home visits, 2 phone calls from the case manager to the dyads, and receiving telephone calls from FCGs during the working hours (Monday through Friday, 9-5). The case manager will target the prioritized risk from the 4 risk areas of FCG problems: depressive symptoms, burden, distress to problematic behaviors of PWDs, and healthy behaviors (Table 1). The intervention mainly consists of 1. needs assessment and nursing education on home environment modification and safety, behavioral management and communication skills(Belle et al., 2006); 2. home-based cognitive stimulation on PWD with simple mathematical practice (Cheng et al., 2013), patient preferred leisure activities (Chiu et al., 2015) and reminiscence by old time photos, stories and toys (Chiu et al., 2013); 3. brief consultation on 4 risk areas related to FCG stress (Belle et al., 2006) and 4. case management to refer the dyads to the hospital-based dementia centers and community resources (Chien et al., 2010). The case manager will assess the recruited dyads at the beginning of the intervention (T0), develop a tailored care plan based on the prioritized risk area of the FCGs and conduct the first home visit in the 1st month to build up a partnership with FCGs, discuss the care plan with the FCGs (and PWDs if possible). Each risk area of each FCG will be dealt with CM components such as education, brief counseling, problem solving and evidence based strategies derived from the Pearlin's theoretical principles. The case manager will teach the FCGs how to implement the home-based cognitive stimulation and cognitive training for PWDs and provide them the daily log for recording these activities and any leisure-time physical activities as well as medical cost. There will be two telephone calls in the 2nd and 3rd months to reinforce the dyads about the taught strategies, collect the log data and remind them the date of the next home visit (4th month). If the problems in each risk area persist until the first phone call, the case manager will discuss this case in a multidisciplinary conference in the participating dementia centers with nurses, social workers, clinical psychologists and neurologists. Then a revised care plan will be developed and additional home visit will be conducted in the 3rd month. If it is necessary, the case manager will refer the dyads to the hospital-based dementia centers, memory clinics or governmental resources. The frequent contacts are to ensure the CM strategies can reflect the changing needs of the FCGs. The definition of compliance is 80% of CM strategies completed by the dyads. The outcome data will be collected after the recruitment in the 4th month (T1), 6th month (T2) and 12th moth (T3) either by home visits or dementia center or memory clinic visits.

To ensure the quality of medical care, both group participants will be followed up at three monthly intervals in the dementia centers. PWDs of the experimental and control groups will receive standard medical treatment as clinically indicated.

For the control group, after the initial assessment, the case manager will give the dyads written information about dementia and its progress as well as home safety during the first home visit. Then case manager will make 2 phone calls in the 2nd and 3rt months for social interactions with the control group and collect the cost data. These phone calls do not involve in active education, consultation or cognitive stimulation and training. The control dyads will remain their usual care, i.e., visiting their primary care physicians or special neurologists for treatments or related consultation as well as education. The participating physicians will be unaware of the dyads allocation to either intervention or control condition. The dyads in the control group have no access to most of the structured and tailored activities. The outcome data will be collected at the 4th month (T1), 6th month (T2) and 12th month (T3)

ELIGIBILITY:
Inclusion Criteria:

1. age being older than 60 years old;
2. having a primary FCG or a secondary FCG who can provides sufficient information and assistant for the PWD; co-residence is not required;
3. PWDs are those with cognitive impairment confirmed by the primary or secondary FCG or participating neurologists

Exclusion Criteria:

1. acute illnesses, impaired sensory symptoms (hearing loss and severe visual problems);
2. acute agitation which requires emergency treatment;
3. chronic alcohol abuse or use of drugs which possibly affect central nervous system functions;
4. presence of major psychiatric disorders within the last 2 years;
5. neurological or systemic illness (e.g. delirium, hypoxia, or unstable thyroid dysfunction);
6. no primary FCG or secondary FCG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The Change of FCG Quality of Life | The outcome data will be collected after the recruitment in the 4th month (T1), 6th month (T2) and 12th moth (T3) either by home visits or dementia center or memory clinic visits.
  The FCG QoL will be measured by the composite score of the measures from the 4 risk areas of FCGs for PWDs using The Center for Epidemiologic Depression (CESD-10), Chinese Caregiving Burden Scale (CBS), Neuropsychological Inventory (NPI) caregiver distress scale, and Health Promotion Profile.

SECONDARY OUTCOMES:
Yielding to FCG role (the PWD status) | The outcome data will be collected after the recruitment in the 4th month (T1), 6th month (T2) and 12th moth (T3) either by home visits or dementia center or memory clinic visits.
  The secondary outcome of the CM intervention is yielding to FCG role based on PWD status: staying at home, admitting to hospital and admitting to nursing home. The time of events and days of staying will be collected through FCGs.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chen Chiu, PhD., Principal Investigator — Chang Gung University
Locations (1):
- Catholic Mercy Hospital, Hukou, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided